CLINICAL TRIAL: NCT04293809
Title: A Phase 1, Pilot, Open Label, Study to Evaluate the Pharmacokinetics, and Safety, of EXPAREL Administered as Pectoral Plane Block in Women Undergoing Breast Augmentation Surgery
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of EXPAREL Administered as a Pectoral Plane Block in Women Undergoing Breast Augmentation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-123
Record Dates: First submitted 2020-02-29; First posted 2020-03-03 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Breast Augmentation
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - EXPAREL (Experimental): A total of 15 subjects will be enrolled in this cohort. Subjects in this cohort will receive 20mL EXPAREL (266mg) with 30mL of saline
  Interventions: Drug: Exparel Injectable Product
- Cohort 2 - EXPAREL (Experimental): A total of 15 subjects will be enrolled. Subjects in this cohort will receive 20mL EXPAREL (266mg) with 30mL of 0.5% bupivacaine HCl (150mg)
  Interventions: Drug: Exparel Injectable Product; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Exparel Injectable Product — bupivacaine liposome injectable suspension
Drug: Bupivacaine Hydrochloride — 1.3%, 13.3 mg/mL
  Arms: Cohort 2 - EXPAREL

SUMMARY:
This is a pilot, open label, single center study in 30 women undergoing breast augmentation. The study will assess and collect information on pharmacokinetics and safety of EXPAREL administered as a pectoral plane block.

A total of 15 subjects will be enrolled in each of the 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or older, undergoing breast augmentation and are American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
2. Able to provide informed consent, adhere to the study schedule, and complete all study assessments
3. Body Mass Index ≥18 and ≤30 kg/m2

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine, NSAIDs)
2. Documented history of long-term diabetes (≥10 years) or severe peripheral vascular disease
3. Renal (serum creatinine level >2mg/dL [176.8 μmol/L]) or hepatic dysfunction (serum alanine or aspartame transferase > 3 times the upper limit of normal)
4. Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post dosing period for pain and which, in the investigator's opinion may confound the post dosing assessments
5. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
6. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
7. Previous participation in an EXPAREL study
8. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the investigator, could interfere with study assessments or compliance
9. Currently pregnant, nursing, or planning to become pregnant during the study
10. Clinically significant medical disease that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other conditions that would constitute a contraindication to participation in the study
11. Currently on neuroleptic agent [e.g., gabapentin, pregabalin (Lyrica), duloxetine (Cymbalta) etc.]
12. Chronic opioid use in the last 30 days (≥30 morphine equivalents/ day)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic 1 (area under the plasma concentration) | predose (up to 15 min before block), 15 min(±10min), 30 min(±5min), and 1(±15min), 2(±15min), 6(±30min), 10(±30min), 18(±1), 26(±1), 36(±2), 48(±2), 60(±2), 72(±3), and 96 (±3) hours from start of study drug administration
  Area under the plasma concentration-versus-time curve (AUC)
Pharmacokinetic 2 (Cmax) | predose (up to 15 min before block), 15 min(±10min), 30 min(±5min), and 1(±15min), 2(±15min), 6(±30min), 10(±30min), 18(±1), 26(±1), 36(±2), 48(±2), 60(±2), 72(±3), and 96 (±3) hours from start of study drug administration
  Maximum plasma concentration
Pharmacokinetic 3 (half-life) | predose (up to 15 min before block), 15 min(±10min), 30 min(±5min), and 1(±15min), 2(±15min), 6(±30min), 10(±30min), 18(±1), 26(±1), 36(±2), 48(±2), 60(±2), 72(±3), and 96 (±3) hours from start of study drug administration
  The apparent terminal elimination half-life (t1/2el)
Pharmacokinetic 4 (apparent clearance) | predose (up to 15 min before block), 15 min(±10min), 30 min(±5min), and 1(±15min), 2(±15min), 6(±30min), 10(±30min), 18(±1), 26(±1), 36(±2), 48(±2), 60(±2), 72(±3), and 96 (±3) hours from start of study drug administration
  Apparent Clearance (CL/F)
Pharmacokinetic 5 (Mean residence time) | predose (up to 15 min before block), 15 min(±10min), 30 min(±5min), and 1(±15min), 2(±15min), 6(±30min), 10(±30min), 18(±1), 26(±1), 36(±2), 48(±2), 60(±2), 72(±3), and 96 (±3) hours from start of study drug administration
  Mean residence time (MRT)

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Nagaraj, MD, PhD, MPH, Study Director — Pacira Pharmaceuticals, Inc
Locations (1):
- HD Research, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: No